CLINICAL TRIAL: NCT05446467
Title: Safety and Efficacy of Pembrolizumab in Combination With Low-dose PF (Cisplatin and 5-Fluorouracil) as Neoadjuvant Treatment for Locally Advanced Head and Neck Squamous Cell Carcinoma: a Multi-center, Single-arm Clinical Study Trial
Brief Title: Pembrolizumab in Combination With Low-dose PFas Neoadjuvant Treatment for Locally Advanced HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Minghua Ge, Director, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KPF20220630
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab+cisplatin + 5-fluorouracil (Experimental): Pembrolizumab+ cisplatin+ 5-fluorouracil+ surgery+ adjuvant treatment+ pembrolizumab maintenance
  Interventions: Combination Product: pembrolizumab+cisplatin + 5-FU

INTERVENTIONS:
Combination Product: pembrolizumab+cisplatin + 5-FU — ivgtt, pembrolizumab 200mg d1+cisplatin20 mg/m2 qd d1-d3 + 5-fluorouracil 3000mg/m2 last for 120hours, six circles. Subjects will undergo surgery after receiving neoadjuvant chemotherapy within 3 weeks, followed by adjuvant therapy and pembrolizumab alone maintenance treatment.

SUMMARY:
A phase Ⅱ open label multi-cencter clinical trail to evaluate the efficacy and safety of pembrolizumab combined with low-dose PF (cisplatin + 5-fluorouracil) in the neoadjuvant treatment of locally advanced head and neck squamous cell carcinoma

DETAILED DESCRIPTION:
The investigatorsdesigned a multi-center, single-arm, small sample clinical pilot study. In the clinical trial, patients were given regimes of induction therapy with PLPF (Pembrolizumab + Low dose- P (Platinum) F (5-Fluorouracil)): 6 cycles of Pembrolizumab treatment. Herein, the investigators describe eight consecutive unselected LA SCCHN (Locally Advanced Head and Neck Squamous Cell Carcinoma) patients based on 6 completed cycles of PLPF induction therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 85 years old
2. Histologically or cytologically proven squamous cell carcinoma of the head and neck; Patients diagnosed with head and neck squamous cell carcinoma with stage III and IV A without distant metastasis according to AJCC staging (8th editon), including squamous cell carcinoma of oropharyngeal (P16-), oral cavity, hypopharyngeal and larynx
3. Measurable primary lesions per RECIST 1.1 criteria
4. Treatment-naive patients without any previous disease-related therapy (except for diagnostic biopsies on primary lesions)
5. ECOG performance status of 0 or 1
6. Selective standard surgery+ standard adjuvant chemo-radiotherapy/radiotherapy as judged by the investigator
7. No active autoimmune disease
8. No concurrent malignancy
9. Life expectancy is estimated to be over 3 months
10. Have sufficient tumour tissue samples available for CPS PD-L1 immunohistochemical examination (22C3 DAKO)
11. No abvious signs of hematological disorders, ANC≥1.5×109 /L, platelets ≥100×109 /L, Hb≥ 90 g/L,WBC ≥3.0×109 /L before enrollment, no blood transfusion and bleeding tendency within 7 days
12. ALT,AST and ALP ≤ 2.5 × upper limit of normal (ULN); Serum bilirubin ≤ 1.5 × ULN, for patients with known Gilbert disease, serum bilirubin ≤ 3 x ULN
13. Serum creatinine ≤1.5 or creatinine clearance>50 mL/min
14. HPV status determined by p16 IHC, in situ hybridization, or by polymerase chain reaction-based assays
15. Able to understand this study, patient and (or) legal representative voluntarily agree to participate in this trial and sign informed consent

Exclusion Criteria:

1. Multiple organs failure
2. HPV p16 positive oropharyngeal cancer
3. Patients with local advanced head and neck squamous cell carcinoma stage T4B and/or N3
4. Patients with distant metastasis
5. Uncontrolled serious diseases that, as assessed by investigator, may affect the subject's treatment with the study protocol, such as serious heart disease, cerebrovascular disease, uncontrolled diabetes mellitus, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.
6. Diagnosis of dementia, altered mental status or any mental illness that would prevent subjects understanding or giving informed consent or completing questionnaires
7. Subjects with ≥ Grade 2 peripheral neuropathy according to CTCAE V5.0
8. Subjects with ≥ Grade 2 hearing impairment according to CTCAE V5.0
9. History of allergy or hypersensitivity to any of the therapeutic ingredients
10. Diagnosis of malignancy within 5 years prior to screening, including HNSCC (other than current HNSCC) and other malignancies; Eligibility is achieved if all of the following criteria are met: malignancies received curative therapy, such as adequately treated cervical carcinoma in situ, non-melanoma cutaneum carcinoma, localized prostate cancer after radical operation, breast ductal carcinoma in situ after radical operation; There was also no evidence of recurrence or metastasis based on imaging and tumor markers
11. Known history of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)
12. Patients diagnosed with nasopharyngeal carcinoma or squamous cell carcinoma whose lesions are located in parts other than the oral cavity, oropharynx, larynx and hypopharynx (such as sinuses, paranasal sinuses and unknown primary site)
13. Participated in other clinical intervention trials or received other investigational therapies within 30 days prior to screening
14. Patients received systemic corticosteroids (prednisone equivalent dose>10mg/day) or other immunosuppressive drugs within 14 days prior to randomization. If there is no active autoimmune disease, inhaled or topical steroid hormones and adrenal hormone replacement therapy with prednisone equivalent doses>10mg per day are permitted
15. Pregnant or breastfeeding; Subjects of childbearing age refuse to accept contraceptive measures
16. Patients unfit for study as assessed by the investigator
17. Received systemic antibiotics within 1 weeks prior to first dose of study therapy or active infection requiring treatment
18. Known history of HBV infection (defined as HBsAg positive) or active HCV infection (defined as HCV RNA detected)
19. Has received live vaccine during study or within 30 days prior to first dose of study therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary site CR rate after neoadjuvant therapy | Up to 6 months
  Measure the primary site CR rate after neoadjuvant therapy

SECONDARY OUTCOMES:
Incidence of adverse reactions during neoadjuvant therapy | up to 2 years
  Incidence of adverse reactions during neoadjuvant therapy
The stages of descent after neoadjuvant therapy | up to 6 months
  The stage of the tumor after neoadjuvant therapy according to the American Joint Committee on Cancer (AJCC) TNM staging system (8th edition) will be evaluated by treating physicians.
Primary site pCR rate after neoadjuvant therapy | Up to 6 months
  Primary site pCR rate after neoadjuvant therapy
EFS | up to 2 years
  EFS is defined as the time from the initial treatment date to the first documented event date, including disease progression, local or distant metastasis as assessed by image or biopsy, or death from any cause, whichever comes first.
DFS | up to 2 years
  DFS is defined as the time from surgery to disease progression or death due to any cause, whichever comes first.
PFS | up to 2 years
  PFS is defined as the time from initial treatment to disease progression or death from any cause, whichever comes first.
OS | 2 years
  OS is defined as the time from initial treatment to death due to any cause.
One year local control rate | up to 6 months
  One year local control rate
1-, 2-year survival rates | up to 2 years
  1-, 2-year survival rates

OTHER OUTCOMES:
Exploratory Outcome2 | Up to 6 months
  Pembrolizumab in combination with low-dose PF (cisplatin + 5-fluorouracil) stratified by CPS PD-L1 status (CPS PD-L1<1, CPS PD-L1>1, and CPS PD-L1 not evaluable/uncertain) ) for the primary CR rate of stage 1 neoadjuvant therapy for locally advanced HNSCC
Exploratory Outcome：biomarkers and single-cell sequencing | up to 2 years
  Immune cell flow analysis, blood MRD detection analysis, single-cell sequencing analysis before and after immune neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Ge, PhD, Principal Investigator — Zhejiang Provincial People's Hospital
Locations (7):
- China (7):
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital School of Medicine,Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - Tianjin Cancer Hospital Airport Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou

IPD SHARING:
Plan to Share IPD: No